CLINICAL TRIAL: NCT00002211
Title: An Open-Label Randomized Study of Delavirdine Mesylate (DLV, Rescriptor) Plus Nelfinavir (NFV), Didanosine (ddI), and Stavudine (d4T) in Triple and Quadruple Treatment Regimens in HIV-1 Infected Individuals
Brief Title: Safety and Effectiveness of Giving Combinations of Three or Four Anti-HIV Drugs to HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmacia and Upjohn (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 228E; 0073
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-04

CONDITIONS: HIV Infections
Keywords: HIV-1; Didanosine; Stavudine; HIV Protease Inhibitors; RNA, Viral; Delavirdine; Reverse Transcriptase Inhibitors; Viral Load; Nelfinavir
MeSH Terms: conditions — HIV Infections | interventions — Nelfinavir; Delavirdine; Stavudine; Didanosine

INTERVENTIONS:
Drug: Nelfinavir mesylate
Drug: Delavirdine mesylate
Drug: Stavudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to see if it is safe and effective to give combinations of three or four anti-HIV drugs to HIV-infected patients. The drugs used in this study are delavirdine (DLV), nelfinavir (NLF), didanosine (ddI), and stavudine (d4T).

DETAILED DESCRIPTION:
This is a multicenter, open-label study. Patients are stratified by HIV-1 RNA levels (20,000 to 200,000 copies/ml and greater than 200,000 copies/ml). Patients are equally randomized to one of four groups and receive antiretroviral therapy for 24 weeks. Group 1 receives delavirdine (DLV) plus nelfinavir (NFV) plus stavudine (d4T). Group 2 receives DLV plus NFV plus didanosine (ddI). Group 3 receives NFV plus d4T plus ddI. Group 4 receives DLV plus NFV plus d4T plus ddI. Patients are evaluated for drug safety and viral burden. Patients may opt to continue on the study for 24 additional weeks, at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are at least 18 years old.
* Are HIV-positive.
* Have a CD4 count of at least 50 cells/mm3.
* Have a viral load of at least 20,000 copies/ml.

Exclusion Criteria

You will not be eligible for this study if you:

* Have taken d4T.
* Have taken protease inhibitors, including NFV.
* Have taken nonnucleoside reverse transcriptase inhibitors.
* Have taken ddI for 1 month or more.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacia & Upjohn, Peapack, New Jersey, United States